CLINICAL TRIAL: NCT04745130
Title: Efficacy and Safety of Sintilimab Combined With Regorafenib and Cetuximab / Sintilimab Combined With Regorafenib in Posterior Line Therapy of Advanced Colorectal Cancer (Regosinti)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rui Liu
Record Dates: First submitted 2021-02-01; First posted 2021-02-09 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Sintilimab, Cetuximab, Regorafenib,Combine,mCRC
Keywords: Sintilimab, Cetuximab, Regorafenib,Combine,mCRC, After the line therapy, curative effect, security

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm 1 (Experimental): KRAS BRAF mutant Sintilimab 200mg D1 Q3W + regafinil 80mg D1-21 Q4W
  Interventions: Drug: KRAS BRAF mutant Sintilimab + regafinil
- Intervention arm 2 (Experimental): KRAS BRAF wild type Sintilimab 200mg d1q3w+ regofinib 80mg d1-21 q4w with cetuximab 500mg/m2 q2w
  Interventions: Drug: Sintilimab，regofinib，cetuximab

INTERVENTIONS:
Drug: Sintilimab，regofinib，cetuximab — KRAS BRAF wild type Sintilimab 200mg d1q3w+ regofinib 80mg d1-21 q4w with cetuximab 500mg/m2 q2w
  Arms: Intervention arm 2
Drug: KRAS BRAF mutant Sintilimab + regafinil — KRAS BRAF mutant Sintilimab 200mg D1 Q3W + regafinil 80mg D1-21 Q4W
  Arms: Intervention arm 1

SUMMARY:
The incidence of colorectal cancer ranks the third in the world and the mortality ranks the second in the world. The incidence and mortality of colorectal cancer have increased in China in the past decade. The incidence of colorectal cancer is associated with dietary patterns, obesity and lifestyle. The 2010 colorectal cancer survey in China showed that the incidence of colorectal cancer was low in the age group below 50 years old, and began to increase rapidly in the age group above 50 years old, reached the maximum in the age group above 70 years old, and decreased after 80 years old.

For advanced colorectal cancer, systemic chemotherapy, local radiotherapy, synchronous or sequential chemoradiotherapy are lack of specificity, killing tumor cells as well as human normal cells, and the space for the traditional cytotoxic chemotherapy drugs to further improve the clinical efficacy of anti-malignant tumor is very limited. Therefore, molecular targeted tumor therapy with strong specificity and relatively small toxic and side effects has gradually become the fourth treatment mode following the three conventional treatment methods of surgery, radiotherapy and chemotherapy. Epidermal growth factor receptor (EGFR) is a clear target for treatment of advanced colorectal cancer. Immunotherapy has been a hot topic in recent years, In the field of colorectal cancer, studies on MSI-H population have been carried out successively since ASCO in 2015.However, the MSI-H population accounts for only 5% of patients with advanced colorectal cancer and 12-15% of total colorectal cancer, and the benefit population is very limited.

Cetuximab is approved for the treatment of advanced colorectal cancer in the United States, Europe and China. Cetuximab in combination with chemotherapy is the standard treatment for RAS wild-type (RAS-WT) colorectal cancer. PD-1 monotherapy has been approved for patients with MSI-H/ DMMR colorectal cancer. The approved PD-1 mAb includes Nivolumab and Pembrolizumab. In some small trials, PD-1 monoclonal antibody combined with Regorafenib showed initial efficacy in patients with MSS type advanced colorectal cancer. EGFR signaling pathway blocker combined with PD-1 antibody, a new treatment mode, is of great significance to enrich the content of immunotherapy for patients with colorectal cancer, improve the survival prognosis of patients, and search for new efficacy predictors.

In conclusion, this study, on the one hand, is expected to confirm that RAS and RAF wild-type advanced colorectal cancer and MSS type can benefit from Sintilimab combined with Regorafenib treatment, and at the same time, observe the effective rate of this regimen in the mutant group, so as to provide reference for clinical selection.

DETAILED DESCRIPTION:
More than 1.8 million new cases of colorectal cancer and 881,000 deaths are expected worldwide in 2018, accounting for about one in 10 cancers, according to the Global Cancer Statistics Report 2018.The incidence of colorectal cancer ranks the third in the world and the mortality ranks the second in the world. The incidence and mortality of colorectal cancer have increased in China in the past decade.The incidence of colorectal cancer is associated with dietary patterns, obesity and lifestyle.

The latest national cancer statistics, "Analysis of Malignant Tumor Epidemiology in China in 2015", showed that the incidence and mortality of colorectal cancer ranked third and fifth in China, respectively. The incidence and mortality of colorectal cancer were both higher in urban areas than in rural areas, and that of males was higher than that of females.In 2010, the incidence of colorectal cancer in China was 26.70/100,000 in urban areas and 15.01/100,000 in rural areas, which was 1.78 times higher than that in rural areas.The top five cities of incidence in China are Shenzhen, Xiamen, Tonghua of Jilin, Guangzhou and Yueyanglou District of Hunan, while the bottom five cities are Hai 'an County of Jiangsu, Tengzhou City of Shandong, Lianshui County of Jiangsu, Tong 'an District of Xiamen and Taixing City of Jiangsu.The 2010 survey of colorectal cancer in China showed that the incidence of colorectal cancer was low in the age group below 50 years old, and began to rise rapidly in the age group above 50 years old, reached the maximum in the age group above 70 years old, and decreased after 80 years old.

For advanced colorectal cancer, with systemic chemotherapy and local radiotherapy, synchronous or sequential radiation and chemotherapy treatment lack of specificity, at the same time of killing tumor cells and normal cells to produce damage effect to human body, and the traditional cytotoxic chemotherapy drugs to further improve the resistance of malignant tumor clinical curative effect of the space is very limited, therefore, strong specificity, side effects of relatively small tumor molecular targeted therapy gradually became the three conventional surgery, radiotherapy and chemotherapy treatment method of the fourth model.Epidermal growth factor receptor (EGFR) is a clear target for treatment of advanced colorectal cancer.Immunotherapy has been a hot topic in recent years.In the field of colorectal cancer, studies on MSI-H population have been carried out successively since ASCO in 2015.However, the MSI-H population accounts for only 5% of patients with advanced colorectal cancer and 12-15% of total colorectal cancer, and the benefit population is very limited.

Clinical studies confirming the third-line treatment of MCRC with cetuximab include Bond, NCICCO.17, etc.The primary objective of the NCICCO.17 study was to investigate the efficacy of cetuximab in patients with advanced colorectal cancer who failed chemotherapy and ceased to receive chemotherapy. It has been confirmed that compared with the best supportive treatment, cetuximab can prolong the survival period of patients and delay the deterioration of quality of life, which is manifested in delaying the deterioration of overall condition and physical function, and has obvious advantages in improving symptoms, highlighting the role of cetuximab in third-line treatment. Cetuximab was approved for second-line treatment of advanced colorectal cancer in the United States and Europe in 2004.Cetuximab combined with irinotecan is the standard second-line treatment for MCRC with oxaliplatin failure. This study included the European BOND study, the MABEL study, the Latin American LABEL study, and the Australian ELSIE study. All patients were tested for EGFR and irinotecan failed. The results showed that the response rate (ORR), disease control rate (DCR), progression-free survival time (PFS) and overall survival time (OS) were similar among different populations, indicating that Cetuximab improved ORR and PFS.Thus, the position of Cetuximab in the second-line treatment of mCRC was consolidated. On September 18, 2019, China's National Medical Products Administration (SFDA) officially approved cetuximab for the first-line treatment of RAS wild-type metastatic colorectal cancer based on the Tailor trial. The Tailor trial compared the efficacy and safety of first-line treatment with cetuximab combined with FOLFOX-4 (5-FU/LV+ oxaliplatin) versus FOLFOX-4 without cetuximab in patients with RAS wild-type metastatic colorectal cancer (MCRC).The primary endpoint was progression-free survival, and secondary endpoints included overall survival, overall response rate, and safety and tolerability. Research into the group of 393 RAS wild-type metastatic colorectal cancer (mCRC) patients with cetuximab combined FOLFOX4 compared with using FOLFOX alone - 4, significantly improve the patient's primary end point, in addition, the secondary endpoint has improved significantly, and well tolerated treatment, no unexpected adverse reaction, good safety and tolerability.

Based on KEYNOTE-016, KEYNOTE-164, and KEYNOTE-028, Pembrolizumab was approved for line 1 and above treatment in patients with MSI-H/ DMMR colorectal cancer, with an ORR of 36%. The CheckMate -142 study was a multi-cohort, phase II study in which Nivolumab was shown to be effective monotherapy in patients with line 2 or higher mSI-H /dMMR colorectal cancer. Phase Ib/II trials of Pembrolizumab in combination with cetuximab for RAS wild-type, EGFR monoclonal antibody primary treatment of advanced or metastatic colorectal cancer confirmed that the two-agent combination was well tolerated. The most common AEs were cutaneous toxicity, hymenopagnesemia, vomiting, and fatigue, and no new AEs occurred.Preliminary results show synergistic effect. PD-1 monotherapy has been approved for the treatment of mSI-H /dMMR patients with colorectal cancer. The approved PD-1 mAb includes Nivolumab and Pembrolizumab.Cetuximab combined with chemotherapy is the standard treatment for RAS wild-type (RAS-WT) colorectal cancer. Phase II clinical trials of Avelumab (PD-L1) in combination with cetuximab and chemotherapy for primary RAS/BRAF wild-type, MSI, or MSS colorectal cancer are ongoing;A phase Ib/II study of Pembrolizumab in combination with cetuximab in patients with RAS-WT metastatic colorectal cancer of line 2 and above is also ongoing. In some small trials, PD-1 monoclonal antibody combined with Regorafenib showed initial efficacy in patients with MSS type advanced colorectal cancer. EGFR signaling pathway blocker combined with PD-1 antibody, a new treatment mode, is of great significance to enrich the content of immunotherapy for patients with colorectal cancer, improve the survival prognosis of patients, and search for new efficacy predictors.

In conclusion, this study, on the one hand, is expected to confirm that RAS and RAF wild-type advanced colorectal cancer and MSS type can benefit from Sintilimab combined with Regorafenib treatment, and at the same time, observe the effective rate of this regimen in the mutant group, so as to provide reference for clinical selection.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old, no gender limitation； 2. Patients with unresectable recurrent or metastatic adenocarcinoma of the colon or rectum, proven histologically or cytologically； 3. Central laboratory tests confirm microsatellite stability (MSS) or microsatellite instability-low (MSI-L) or proficiency of MMR (PMMR)； 4. For patients who have previously failed systemic therapy for relapsed or metastatic colorectal cancer, or who are intolerant to treatment, the time for disease progression after the last systemic therapy should not exceed 3 months。Systemic therapy must contain two or more of fluorouracil, oxaliplatin, and irinotecan, and may include or not targeted therapy (bevacizumab, cetuximab, etc.)； 5. Patients must have a measurable disease (RECIST v1.1)；

  1. Non-lymph node lesions with the longest single diameter ≥10mm, or lymph node lesions with short diameter ≥15mm；
  2. Lesion after previous local treatment, such as radiotherapy or ablation, can also be a measurable target if it has been clearly developed according to RECIST 1.1 and the longest single diameter is ≥10mm。 6．ECOG PS：0-1； 7．Life expectancy of more than 3 months； 8. Good organ function (no blood transfusion, no use of hematopoietic stimulating factor, no albumin or blood products within 14 days prior to examination)；

  <!-- -->

  1. platelets(PLT)≥75,000 /mm3；
  2. Absolute neutrophil(ANC)≥1,500 /mm3；
  3. hemoglobin(Hb)≥9.0 g/dl；
  4. international normalized ratio(INR)≤1.5；
  5. Total bilirubin ≤2 times the institutional upper limit of normal (ULN)；
  6. Aspartate aminotransferase(AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase(ALT)(serum glutamate pyruvate transaminase [SPGT])≤3X institutional ULN (or≤5 times ULN in case of liver metastasis)；
  7. Creatinine(Cr)≤1.5×ULN and creatinine clearance(CrCl)≥60mL/min； 9. Use contraception and avoid breast-feeding during the study period and for 3 months after the last dosing;Male subjects must agree to use contraception for the duration of the study and for 3 months after the last dosing； 10. Able to understand and willing to sign written informed consent。

Exclusion Criteria:

* 1. Study any other malignancy with a primary site or histological type different from that of CRC that was diagnosed within 5 years prior to treatment initiation, other than adequately treated basal or squamous cell skin cancer or cervical carcinoma in situ； 2. Central laboratory tests confirm microsatellite instability-high(MSI-H) or DNA mismatch repair defcient (dMMR)； 3. Previous treatment with Regorafenib, PD-1/PD-L1/PD-L2 antibodies, or other co-stimulatory targets or checkpoints on T cells； 4. Known to be allergic to the study drug or excipient, or to similar drugs； 5. Known allergy to the study drug or excipient, or to similar drugs received immunosuppressive drugs within 2 weeks prior to the commencement of study treatment (excluding inhaled corticosteroids or other systemic steroids ≤10 mg/ day of prednisone or equivalent pharmacological dose)； 6. A live attenuated vaccine was scheduled to be given 4 weeks before the start of study treatment or during the study period； 7. CYP3A4 inducers or inhibitors should not be discontinued 1 week before and during study treatment； 8. Central nervous system metastases are known to occur； 9. Any autoimmune disease or history of autoimmune disease； 10. Presenting any autoimmune disease or unwell controlled hypertension with a history of autoimmune disease (SBP ≥140 mmHg or Diastolic BP ≥90 mmHg)； 11. Clear bleeding tendency, hemoptysis, hematemesis and stool。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 2 years
  Overall Survival (OS) (median) was determined using the number of months measured from the initial date of treatment to the recorded date of death of participants.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | up to 6 months
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Objective Response Rate | Up to 12months
  The objective response rate is estimated by the proportion (percentage) of participants with the best response of complete response (CR), or partial response (PR) by RECIST 1.1 criteria, with corresponding exact 95% confidence limits being reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Rui Liu, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes